CLINICAL TRIAL: NCT04778917
Title: Observation and Treatment of Pulmonary Microthrombosis in Childhood Pneumonia With Elevated D-dimer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Institute of Pediatrics, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W12-1
Record Dates: First submitted 2020-03-19; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Pneumonia
Keywords: D-dimer,pneumonia,children
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Small dose low molecular weight heparin (Experimental): Low molecular weight heparin calcium 100 units / kg/day, subcutaneous injection, 5-10 days of treatment or D-dimer recovery normal.
  Interventions: Drug: Low-Molecular-Weight Heparins Calcium Injection
- High dose of low molecular weight heparin (Experimental): low molecular weight heparin calcium 200 units /kg/day, subcutaneous injection, treatment for 7 days or D-dimer return to normal.
  Interventions: Drug: Low-Molecular-Weight Heparins Calcium Injection
- Vacuity contrast group (Placebo Comparator): Conventional treatment for children with pneumonia, without the use of low molecular weight heparin.
  Interventions: Drug: Low-Molecular-Weight Heparins Calcium Injection
- contrast group (No Intervention): Conventional treatment for children with pneumonia, without the use of low molecular weight heparin.

INTERVENTIONS:
Drug: Low-Molecular-Weight Heparins Calcium Injection — We use different dose of low-molecular-weight heparins calcium injection to different interventions
  Arms: High dose of low molecular weight heparin; Small dose low molecular weight heparin; Vacuity contrast group

SUMMARY:
Objective

1. Master the clinical feathers, imaging features and laboratory diagnosis characteristics and economic costs of children pneumonia with higher D-dimer:

1. Compare the characteristics of different groups of children in the course of the disease，clinicalsymptoms and signs;
2. All the children in the study need to do enhanced CT, to observe if there were intrapulmonary vascular thrombosis and necrosis pneumonia signs;
3. compared changes of coagulation index beside D-dimer.

2. Compared with low molecular weight heparin prevention Disseminated intravascular coagulation（DIC） dose and instructions to the recommended dose in safety and effectiveness,and proposed elevated anticoagulation D-Dimer specification of the clinical treatment of children with pneumonia.

Background and rationale:

Pneumonia is the main cause of lung function injury and death in children. The high blood coagulation state can lead to the formation of pulmonary vascular thrombosis, local pulmonary ischemia and necrosis, which may be an important mechanism for the occurrence of necrotizing pneumonia and pulmonary embolism in children with pneumonia. Elevated D-dimer is an important predictor of pulmonary thrombosis and necrotizing pneumonia. At present, D-Dimer in many children with severe pneumonia is found to increase, the symptom is severe, the late stage of the performance of necrotizing pneumonia, seriously affect the children's lung function and quality of life.

DETAILED DESCRIPTION:
This is a randomized, controlled, single blind trial(Researchers are not blind, patients are blind).

1.Patient population

1. .Experience group We will recruit 93 cases in our trial.All of them are with simple pneumonia and are hospitalized in the respiratory department of our hospital, also D-dimer is higher than or equal to 500ug / L, 93 cases as the observation group, were randomly divided into A, B, C three sub group.
2. .Control group We will recruit 31 cases in our control group.And children in this group are also with simple pneumonia,they will be similar with the experience group children at the age, the disease course but their D-Dimer is lower than 500 ug/L.

2.Randomized methods: A random number table was created by the statistical staff of the non-present research group using SAS to generate random numbers table before the start of the study. Selected children are in accordance with the A, B, C three groups of 1:1:1 ratio distribution.

3.Study method: Fasting venous blood was extracted from all the children from the second morning after admission to complete the coagulation function, blood routine, biochemical and related inflammatory indicators and complete chest CT examination。The above indicators were monitored dynamically during hospitalization.

4.Study protocal:

Study group:

Group A :Conventional treatment for children with pneumonia, without the use of low molecular weight heparin.

Group B :Group B with prevention of DIC amount: low molecular weight heparin calcium 50-100 units / kg, once or twice subcutaneous injection, 5-10 days of treatment or D-Dimer recovery normal. According to Huang Ke, disseminated intravascular coagulation, Huang Shaoliang, Zhou Dunhua, editor in chief of pediatric hematology clinical manual, Third Edition, 601-602.

Group C :Group C with anticoagulant therapy: low molecular weight heparin calcium 100 units /kg, subcutaneous injection, two times a day, treatment for 7 days orD-Dimer return to normal. Low molecular weight heparin calcium.

Control group :Conventional treatment for children with pneumonia, without the use of low molecular weight heparin.

5.Statistical methods

Statistical analysis system(SAS).2 software was used for statistical analysis . The continuous variables of the central tendency and the discrete trend are represented by the median and the four point spacing, and the categorical variables are described by the constituent ratio. Normal distribution of continuous variables between the 22 comparison using T test, multiple comparisons using ANOVA. Non normal distribution of continuous variables between the 22 comparison using Rank Sum Test Wilcoxon, multiple comparisons using Kruskal-Wallis method. Statistical testing methods used properly. All the tests were taken by alpha =0.05.

6.Study objection:

1. .Compare the group A with the control group of the clinical features
2. . Compare all of the patients in the observation group with the control group of the chest CT features
3. .To observe the efficacy and safety of anticoagulant therapy to children with D-dimer increased pneumonia

7.Sample size estimation：

As there is no evaluation of the efficacy of children with pneumonia combined with elevated D-Dimer in China, studies have shown that severe pneumonia is often accompanied by elevated D-Dimer. Therefore, this study only estimates the sample size based on the effective rate of heparin in the treatment of severe pneumonia. According to Wang Xuanzhu's research [Wang Xuanzhu. The efficacy of heparin in the treatment of severe pneumonia in children and its effect on platelet parameters and D-dimers], the effective rate of conventional methods in the treatment of severe pneumonia is 76.6%, and the effective rate of low-dose heparin treatment is 95.8%. This study adopts a two-sided test, taking α=0.05, β=0.20, u0.05/2=1.96, u0.2=0.8, p1=0.766, p2=0.958.Considering the possible loss to follow-up rate in this study is 10%, the sample size of each group should be: 31.

8. Reporting for adverse events

Liver function, coagulation function, and platelet monitoring were performed for each child in the group. If there is a tendency to bleeding, the test was immediately terminated and corresponding treatment was given.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of simple pneumonia
* Age 28 days to 18 years

Exclusion Criteria:

* With congenital heart disease
* With kidney disease
* With blood system diseases
* With paralysis
* With muscle tension
* With fracture,
* With a family history of thrombotic disease
* With indwelling central venous catheters
* With parenteral nutrition, neoplastic disease
* With primary immunodeficiency disease

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Lung imaging absorption improvement time after treatment | Change from basline in lung imaging at 1 month
  The enrolled children were subjected to weekly imaging examinations to determine the time for the absorption of lung inflammation to improve.Criteria for evaluating the severity of CT changes (large lung shadows or dot shadows in CT images) : Criteria for improvement of lung imaging absorption: no obvious lesion absorption, no absorption or large patchy shadow; Partial absorption of lesions: there is absorption, but there is still patchy shadow or cloud flocculent shadow; Obvious absorption of lesions: no abnormalities or only a little light in the lung.
Time to improve cough symptoms | 2 weeks
  The clinician will judge the improvement time of the child's cough symptoms
Heat retreat time | 2 weeks
  The time required for temperature to drop below 37.3℃ after treatment.
The time to disappear rhonchus in the lungs | 2 weeks
  The clinician will judge the absorption time of dry and wet rhonchus in the lungs.

SECONDARY OUTCOMES:
Average hospital stay time | 2weeks to 4weeks
  The time required from the child's admission to the improvement and discharge
The degree of coagulation improvement | 2 weeks
  Laboratory test indicators include: platelet count (PLT), prothrombin time, partial thromboplastin time Prothrombin time（PT）\Activated partial thromboplastin time（APTT）, protein fiber, fiber protein degradation product Fibrinogen（FIB）\Fibrinogen degradation products（FDP）, D-dimer, Antithrombin III（AT-III）.Compare the improvement degree of the above indicators in each group before and after treatment.
Differences in inflammation indicators in each group | basline
  The inflammatory markers included CRP, ESR and WBC counts.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Cao, MD, Principal Investigator — Capital Institute of Pediatrics, China
Locations (1):
- Capital Institute of Pediatrics, Beijing, China

REFERENCES:
- [Background] Esposito S, Cohen R, Domingo JD, Pecurariu OF, Greenberg D, Heininger U, Knuf M, Lutsar I, Principi N, Rodrigues F, Sharland M, Spoulou V, Syrogiannopoulos GA, Usonis V, Vergison A, Schaad UB. Antibiotic therapy for pediatric community-acquired pneumonia: do we know when, what and for how long to treat? Pediatr Infect Dis J. 2012 Jun;31(6):e78-85. doi: 10.1097/INF.0b013e318255dc5b. PMID 22466326
- [Background] Schroeder JD, McKenzie AS, Zach JA, Wilson CG, Curran-Everett D, Stinson DS, Newell JD Jr, Lynch DA. Relationships between airflow obstruction and quantitative CT measurements of emphysema, air trapping, and airways in subjects with and without chronic obstructive pulmonary disease. AJR Am J Roentgenol. 2013 Sep;201(3):W460-70. doi: 10.2214/AJR.12.10102. PMID 23971478
- [Background] Litmanovich DE, Hartwick K, Silva M, Bankier AA. Multidetector computed tomographic imaging in chronic obstructive pulmonary disease: emphysema and airways assessment. Radiol Clin North Am. 2014 Jan;52(1):137-54. doi: 10.1016/j.rcl.2013.09.002. PMID 24267715
- [Background] Youn YS, Lee KY, Hwang JY, Rhim JW, Kang JH, Lee JS, Kim JC. Difference of clinical features in childhood Mycoplasma pneumoniae pneumonia. BMC Pediatr. 2010 Jul 6;10:48. doi: 10.1186/1471-2431-10-48. PMID 20604923
- [Background] Madzhuga AV, Somonova OV, Elizarova AL, Sviridova SP, Zubrikhin GN. [The clinical value of D-dimer in the diagnosis and treatment of thromboembolic complications and DIC syndrome in cancer patients]. Anesteziol Reanimatol. 2005 Sep-Oct;(5):55-7. Russian. PMID 16318055
- [Background] Zhao D, Ding R, Mao Y, Wang L, Zhang Z, Ma X. Heparin rescues sepsis-associated acute lung injury and lethality through the suppression of inflammatory responses. Inflammation. 2012 Dec;35(6):1825-32. doi: 10.1007/s10753-012-9503-0. PMID 22782595
- [Background] Lankisch P, Laws HJ, Wingen AM, Borkhardt A, Niehues T, Neubert J. Association of nephrotic syndrome with immune reconstitution inflammatory syndrome. Pediatr Nephrol. 2012 Apr;27(4):667-9. doi: 10.1007/s00467-011-2069-5. Epub 2011 Dec 29. PMID 22203364
- [Background] van der Poll T, de Boer JD, Levi M. The effect of inflammation on coagulation and vice versa. Curr Opin Infect Dis. 2011 Jun;24(3):273-8. doi: 10.1097/QCO.0b013e328344c078. PMID 21330919